CLINICAL TRIAL: NCT03499353
Title: A PHASE 2, NON RANDOMIZED, OPEN LABEL, SINGLE ARM, MULTI CENTER STUDY OF TALAZOPARIB FOR NEOADJUVANT TREATMENT OF GERMLINE BRCA1/2 MUTATION PATIENTS WITH EARLY HUMAN EPIDERMAL GROWTH FACTOR RECEPTOR 2 NEGATIVE BREAST CANCER
Brief Title: Talazoparib For Neoadjuvant Treatment Of Germline BRCA1/2 Mutation Patients With Early Human Epidermal Growth Factor Receptor 2 Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated based on Pfizer's change in clinical development strategy not related to safety and efficacy.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3441020; TALAZOPARIB NEOADJ BC (Other: Alias Study Number)
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Early Breast Cancer
Keywords: Neoadjuvant Therapy, HUMAN EPIDERMAL GROWTH FACTOR RECEPTOR 2 NEGATIVE Breast Cancer, BRCA Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Intervention Model Description: THIS IS AN OPEN LABEL SINGLE ARM STUDY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TALAZOPARIB (Experimental): SINGLE ARM, NON-RANDOMIZED
  Interventions: Drug: TALAZOPARIB

INTERVENTIONS:
Drug: TALAZOPARIB — Talazoparib 1mg/day

SUMMARY:
A PHASE 2, NON RANDOMIZED, OPEN LABEL, SINGLE ARM, MULTI CENTER STUDY OF TALAZOPARIB FOR NEOADJUVANT TREATMENT OF GERMLINE BRCA1/2 MUTATION PATIENTS WITH EARLY HUMAN EPIDERMAL GROWTH FACTOR RECEPTOR 2 NEGATIVE BREAST CANCER

DETAILED DESCRIPTION:
TALAZOPARIB (PARP INHIBITOR) FOR NEOADJUVANT TREATMENT OF GERMLINE BRCA1/2 MUTATION PATIENTS WITH EARLY HUMAN EPIDERMAL GROWTH FACTOR RECEPTOR 2 NEGATIVE BREAST CANCER. THIS IS A MONOTHERAPY TREATMENT FOR 24 WKS FOLLOWED BY SURGERY TO EVALUATE PATHOLOGICAL COMPLETE RESPONSE.

ELIGIBILITY:
Inclusion Criteria:

* Germline BRCA 1/2 Mutation Positive
* Women and men at least 18 years of age or older.
* Histologically confirmed invasive adenocarcinoma of the breast
* HER2 negative breast cancer as defined by ASCO-CAP criteria
* Tumor greater than or equal toT1, N0-3
* No evidence of distant metastasis
* Adequate bone marrow, hepatic, and renal function
* ECOG performance status 0 or 1

Exclusion Criteria:

* Any other previous antitumor therapies for the current cancer event. Treatment for ductal carcinoma in situ (DCIS) is allowed; ie, surgery, hormonal therapy and radiation.
* Evidence of distant metastasis apparent prior to randomization
* Patients with inflammatory breast carcinoma
* Malignancy within the last 3 years, except: Stage 1 melanoma which does not require any further treatment after adequate surgical excision; adequately treated non melanoma skin cancer; Curatively treated in situ cancer of the cervix; Stage 1, Grade 1 endometrial carcinoma; or Adequately treated contralateral breast carcinoma which has been disease free for a year; Other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for 5 years.
* Previous or concomitant systemic anti cancer therapies used for the treatment of cancer in the last 3 years.
* Prior treatment with a PARP inhibitor in any disease setting
* Concomitant use of Strong P gp inhibitors or inducers or BCRP inhibitors
* Patients who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol
* Major surgery within 14 days prior to study entry
* Known history of cardiac disease, for example : Myocardial infarction or symptomatic cardiac ischemia within 24 weeks before screening; Congestive heart failure New York Heart Association Class III or IV; History of clinically significant ventricular arrhythmias within one year prior to randomization; History of Mobitz II second degree or third degree heart block, uncontrolled hypertension.
* Active clinically significant infection
* Clinically significant bleeding diathesis or coagulopathy
* Non healing wound, ulcer or bone fracture
* Known hypersensitivity to any of the components of talazoparib
* Patients with myelodysplastic syndrome/acute myeloid leukemia
* Patients with uncontrolled seizures.
* Any evidence of other disease or any concomitant medical or psychiatric problems which in the opinion of the Investigator would prevent completion of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (93):
- United States (93):
  - Banner Gateway Medical Center, Gilbert, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - PMK Medical Group Inc., dba Ventura County Hematology Oncology Specialists, Camarillo, California
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - City of Hope Investigational Drug Services (IDS), Duarte, California
  - The Oncology Institute of Hope & Innovation, Glendale, California
  - Glendale Adventist Medical Center, Glendale, California
  - The Oncology Institute of Hope & Innovation, Long Beach, California
  - UC Irvine Health, Orange, California
  - UC Irvine Medical Center, Orange, California
  - PMK Medical Group Inc., dba Ventura County Hematology Oncology Specialists, Oxnard, California
  - Emad Ibrahim, MD, INC., Redlands, California
  - The Oncology Institute of Hope & Innovation, Santa Ana, California
  - Stanford Cancer Institute, Stanford, California
  - Stanford Hospital and Clinics, Stanford, California
  - Stanford Women's Cancer Center, Stanford, California
  - PMK Medical Group Inc., dba Ventura County Hematology Oncology Specialists, Ventura, California
  - The Oncology Institute of Hope & Innovation, West Covina, California
  - The Oncology Institute of Hope & Innovation, Whittier, California
  - ICRI, Whittier, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Englewood, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Innovative Medical Research of South Florida, Inc, Aventura, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Rush University Medical Center, Professional Office Building Infusion Pharmacy, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Rush Oak Park Hospital, Oak Park, Illinois
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Summit Medical Group PA, Florham Park, New Jersey
  - St. Luke's Hospital - Warren Campus, Phillipsburg, New Jersey
  - St. Luke's Warren Physician Group, Phillipsburg, New Jersey
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - St. Luke's Hematology Oncology Specialists, Allentown, Pennsylvania
  - St. Luke's Hospital - Allentown Campus, Allentown, Pennsylvania
  - St. Luke's Hematology Oncology Specialists, Bethlehem, Pennsylvania
  - St. Luke's Hospital - Bethlehem Campus, Bethlehem, Pennsylvania
  - St. Luke's Hospital - Miners Campus, Coaldale, Pennsylvania
  - St Luke's Hospital - Anderson Campus, Easton, Pennsylvania
  - St. Luke's Hospital - Anderson Campus, Easton, Pennsylvania
  - UPMC Hillman Cancer Center Mountainview Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Cancer Centers East Oxford Drive, Monroeville, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center North Hills at Passavant, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center UPMC Passavant, Pittsburgh, Pennsylvania
  - St. Luke's Hospital - Quakertown Campus, Quakertown, Pennsylvania
  - St. Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Uniontown, Uniontown, Pennsylvania
  - UPMC Hillman Cancer Center Washington, Washington, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera Specialty Hospital, Sioux Falls, South Dakota
  - Brig Center for Cancer Care and Survivorship, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Texas Oncology - Allen, Allen, Texas
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - U.T. MD Anderson Cancer Center, Investigational Pharmacy Services - Unit 376, Houston, Texas
  - U.T. MD Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology - Round Rock, Round Rock, Texas
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - UW Health University Hospital - Pharmaceutical Research Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Litton JK, Beck JT, Jones JM, Andersen J, Blum JL, Mina LA, Brig R, Danso M, Yuan Y, Abbattista A, Noonan K, Niyazov A, Chakrabarti J, Czibere A, Symmans WF, Telli ML. Neoadjuvant Talazoparib in Patients With Germline BRCA1/2 Mutation-Positive, Early-Stage Triple-Negative Breast Cancer: Results of a Phase II Study. Oncologist. 2023 Oct 3;28(10):845-855. doi: 10.1093/oncolo/oyad139. PMID 37318349
- [Derived] Litton JK, Scoggins ME, Hess KR, Adrada BE, Murthy RK, Damodaran S, DeSnyder SM, Brewster AM, Barcenas CH, Valero V, Whitman GJ, Schwartz-Gomez J, Mittendorf EA, Thompson AM, Helgason T, Ibrahim N, Piwnica-Worms H, Moulder SL, Arun BK. Neoadjuvant Talazoparib for Patients With Operable Breast Cancer With a Germline BRCA Pathogenic Variant. J Clin Oncol. 2020 Feb 10;38(5):388-394. doi: 10.1200/JCO.19.01304. Epub 2019 Aug 28. PMID 31461380
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441020

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 61 participants were enrolled and treated with talazoparib.
Groups:
- Talazoparib 1 mg QD: During talazoparib treatment period, participants received oral administration of talazoparib 1 mg once daily (QD) for 24 weeks (6 cycles, 4 weeks per cycle), or 0.75 mg QD in case of moderate renal impairment at baseline, followed by definitive breast surgery within a maximum of 6 weeks of last dose.
  Safety follow-up (end of treatment visit) occurred approximately 28 calendar days after the last dose of talazoparib or after permanent treatment discontinuation or before initiation of a new antineoplastic therapy (whichever occurred first).
  Long-term follow-up was planned to be at least 3 years, which started from the date of surgery for event-free survival (EFS) and after first dose of talazoparib for overall survival (OS).
Period: Treatment
Arm/Group | Talazoparib 1 mg QD
Started | 61
Completed | 45
Not Completed | 16
Not completed — Adverse Event | 3
Not completed — Progressive Disease | 10
Not completed — Other | 1
Not completed — Withdrawal by Subject | 2
Period: Safety Follow-up
Arm/Group | Talazoparib 1 mg QD
Started | 49
Received Treatment | 0
Completed | 49
Not Completed | 0
Period: Long-Term Follow-up
Arm/Group | Talazoparib 1 mg QD
Started | 58
Received Treatment | 0
Completed | 0
Not Completed | 58
Not completed — Death | 2
Not completed — Study Terminated By Sponsor | 55
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received any amount of talazoparib.
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 44.6 (12.7)
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 37
  45-64 Years | 18
  >=65 Years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47
  Black or African American | 7
  Asian | 3
  Not reported | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 1
  African American | 7
  Ashkenazi Jew | 1
  Other | 49
  Not reported | 3
Number of Participants with Triple Negative Breast Cancer (TNBC) at Baseline [Count of Participants; unit: Participants] — Participants with TNBC at baseline were defined as participants that lacked estrogen receptor (ER Negative), progesterone receptor (PR Negative) and human epidermal growth factor receptor 2 (HER2 Negative) at baseline.
  Participants | 61
Duration of Breast Cancer at Baseline [Median (Full Range); unit: Weeks] — Duration (since onset) was defined as time (weeks) from histopathological (primary) diagnosis until study entry (baseline).
  Weeks | 3.57 [0.43 to 21.14]
Number of Participants with Breast Cancer Gene 1/2 (BRCA1/2) Mutations at Baseline [Count of Participants; unit: Participants] — Participants with BRCA1/2 mutations at baseline were defined as participants with positive Myriad BRCA1/2 laboratory test results at baseline.
  Participants
    BRCA1 | 48
    BRCA2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Pathological Complete Response (pCR) as Per Independent Central Review (ICR) in Evaluable Analysis Set as Per ICR With 80% Confidence Interval (CI)
Description: pCR was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (ie, ypT0/Tis ypN0 in the current American Joint Committee on Cancer [AJCC] staging system). pCR rate by ICR was defined as the percentage of participants achieving pCR by ICR after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the evaluable population (Evaluable Analysis Set as per ICR). The exact CI was calculated using the Blaker's method.
Time Frame: Date of surgery (maximum of approximately 8 months post-baseline) (assessed within a maximum of 6 weeks of last dose of talazoparib)
Population: The analysis population included all participants enrolled who received at least 80% of the dose of talazoparib prescribed at treatment start (1 mg/day, with the exception of participants with baseline moderate renal impairment who received a starting dose of 0.75 mg/day) and underwent breast surgery and pCR assessment by ICR, as well as participants who progressed or died before pCR could be assessed by ICR (these participants were considered as non-responders).
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 48
Percentage of participants | 45.8 [36.42 to 55.22]

2. Primary Outcome: Percentage of Participants Achieving pCR as Per ICR in Evaluable Analysis Set as Per ICR With 95% CI
Description: pCR was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (ie, ypT0/Tis ypN0 in the current AJCC staging system). pCR rate by ICR was defined as the percentage of participants achieving pCR by ICR after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the evaluable population (Evaluable Analysis Set as per ICR). The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 48
Percentage of participants | 45.8 [31.98 to 60.62]

3. Secondary Outcome: Percentage of Participants Achieving pCR as Per ICR in Intention-to-Treat (ITT) Analysis Set With 80% CI
Description: pCR was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (ie, ypT0/Tis ypN0 in the current AJCC staging system). pCR rate by ICR in ITT Analysis Set was defined as the percentage of participants achieving pCR by ICR after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the ITT Analysis Set. The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Percentage of participants | 49.2 [40.97 to 57.39]

4. Secondary Outcome: Percentage of Participants Achieving pCR as Per ICR in ITT Analysis Set With 95% CI
Description: as for outcome 3
Time Frame: as for outcome 1
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Percentage of participants | 49.2 [36.70 to 61.63]

5. Secondary Outcome: Percentage of Participants Achieving pCR as Per Investigator in Evaluable Analysis Set as Per Investigator
Description: pCR was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (ie, ypT0/Tis ypN0 in the current AJCC staging system). pCR rate by investigator was defined as the percentage of participants achieving pCR by investigator review after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the evaluable population (Evaluable Analysis Set as per Investigator). The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: The analysis population included all participants enrolled who received at least 80% of the talazoparib dose prescribed at treatment start (1 mg/day, except participants with baseline moderate renal impairment who received a starting dose of 0.75 mg/day) and underwent breast surgery and pCR assessment by investigator, as well as participants who progressed or died before pCR could be assessed by investigator (these participants were considered as non-responders).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 48
Percentage of participants | 45.8 [31.98 to 60.62]

6. Secondary Outcome: Percentage of Participants Achieving pCR as Per Investigator in ITT Analysis Set
Description: pCR was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (ie, ypT0/Tis ypN0 in the current AJCC staging system). pCR rate by investigator in ITT Analysis Set was defined as the percentage of participants achieving pCR by investigator review after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the ITT Analysis Set. The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Percentage of participants | 47.5 [35.03 to 60.09]

7. Secondary Outcome: Percentage of Participants Achieving pCR in Breast Only as Per Investigator in Evaluable Analysis Set as Per Investigator
Description: pCR in breast was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen following completion of neoadjuvant therapy with talazoparib. pCR rate in breast by investigator was defined as the percentage of participants achieving pCR in breast by investigator review after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the evaluable population (Evaluable Analysis Set as per Investigator). The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 48
Percentage of participants | 45.8 [31.98 to 60.62]

8. Secondary Outcome: Percentage of Participants Achieving pCR in Breast Only as Per Investigator in ITT Analysis Set
Description: pCR in breast was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen following completion of neoadjuvant therapy with talazoparib. pCR rate in breast by investigator in ITT Analysis Set was defined as the percentage of participants achieving pCR in breast by investigator review after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the ITT Analysis Set. The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Percentage of participants | 47.5 [35.03 to 60.09]

9. Secondary Outcome: Percentage of Participants Achieving pCR in Breast Only as Per ICR in Evaluable Analysis Set as Per ICR
Description: pCR in breast was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen following completion of neoadjuvant therapy with talazoparib. pCR rate in breast by ICR was defined as the percentage of participants achieving pCR in breast by ICR after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the evaluable population (Evaluable Analysis Set as per ICR). The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 48
Percentage of participants | 47.9 [34.11 to 62.75]

10. Secondary Outcome: Percentage of Participants Achieving pCR in Breast Only as Per ICR in ITT Analysis Set
Description: pCR in breast was defined as the absence of residual invasive cancer in the breast and axillary lymph nodes on hematoxylin and eosin evaluation of the complete resected breast specimen following completion of neoadjuvant therapy with talazoparib. pCR rate in breast by ICR in ITT Analysis Set was defined as the percentage of participants achieving pCR in breast by ICR after talazoparib treatment for 24 weeks, followed by surgery, among all participants in the ITT Analysis Set. The exact CI was calculated using the Blaker's method.
Time Frame: as for outcome 1
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Percentage of participants | 50.8 [38.37 to 63.30]

11. Secondary Outcome: Percentage of Participants With Residual Cander Burden (RCB) as Per ICR in Evaluable Analysis Set as Per ICR
Description: The RCB is a continuous index derived from the following: primary tumor dimensions; cellularity of the tumor bed; axillary nodal burden. Residual cancer burden by ICR is reported as a categorical variable with four classes (categories): RCB 0 (pCR), I (minimal RCB), II (moderate RCB), III (extensive RCB). Participants who had progressive disease or was unable to be assessed for RCB due to missing required axillary specimen were counted in the "Missing" category. The simultaneous exact CI was calculated using Goodman's method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 48
Percentage of participants
  RCB - 0 | 45.8 [29.0 to 63.7]
  RCB - I | 0.0 [0.0 to 12.1]
  RCB - II | 31.3 [17.2 to 49.8]
  RCB - III | 0.0 [0.0 to 12.1]
  Missing (Participants who had progressive disease or with missing required axillary specimen) | 22.9 [11.2 to 41.2]

12. Secondary Outcome: Percentage of Participants With RCB as Per ICR in ITT Analysis Set
Description: as for outcome 11
Time Frame: as for outcome 1
Population: The analysis population included all participants who received any amount of talazoparib
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Percentage of participants
  RCB - 0 | 49.2 [33.6 to 64.9]
  RCB - I | 1.6 [0.2 to 12.6]
  RCB - II | 27.9 [15.8 to 44.2]
  RCB - III | 0.0 [0.0 to 9.8]
  Missing (Participants who had progressive disease or with missing required axillary specimen) | 21.3 [11.0 to 37.3]

13. Secondary Outcome: Probability of Being Event-Free at 3 Years in Evaluable Analysis Set
Description: Event-Free Survival (EFS) is defined as the time from surgery date to first documentation of local or distant recurrence or death or initiation of antineoplastic therapy before documentation of first relapse. Participants discontinuing study before documentation of first relapse or death, but after surgery were censored observations for EFS. EFS at 3 years is defined as the probability of being event free at 3 years after surgery using Kaplan Meier methods.
Time Frame: 3 years after surgery
Population: The analysis population included all participants enrolled who received at least 80% of the dose prescribed at treatment start (1 mg/day, except those with baseline moderate renal impairment who received a starting dose of 0.75 mg/day) and underwent breast surgery and pCR assessment, and participants who progressed or died before pCR could be assessed. EFS at 3 years was not analyzed as the 3-year threshold was not reached at study termination, therefore number of participants analyzed was 0.
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 0

14. Secondary Outcome: Probability of Being Alive at 3 Years in Evaluable Analysis Set
Description: Overall Survival (OS) is defined as the time from first dose of talazoparib to death due to any cause. Participants not known to have died at the time of the analysis were right censored on the date they were last known to be alive before the analysis data cutoff date. OS at 3 years is defined as the probability of being alive at 3 years after first dose of talazoparib using Kaplan Meier methods.
Time Frame: 3 years after first dose of talazoparib
Population: The analysis population included all participants enrolled who received at least 80% of the dose prescribed at treatment start (1 mg/day, except those with baseline moderate renal impairment who received a starting dose of 0.75 mg/day) and underwent breast surgery and pCR assessment, and participants who progressed or died before pCR could be assessed. OS at 3 years was not analyzed as the 3-year threshold was not reached at study termination, therefore number of participants analyzed was 0.
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 0

15. Secondary Outcome: Probability of Being Alive at 3 Years in ITT Analysis Set
Description: OS is defined as the time from first dose of talazoparib to death due to any cause. Participants not known to have died at the time of the analysis were right censored on the date they were last known to be alive before the analysis data cutoff date. OS at 3 years is defined as the probability of being alive at 3 years after first dose of talazoparib using Kaplan Meier methods.
Time Frame: 3 years after first dose of talazoparib
Population: The analysis population included all participants who received any amount of talazoparib. OS at 3 years was not analyzed as no participants had yet reached the 3-year threshold when the study was terminated, therefore the number of participants analyzed for this outcome measure was 0.
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs that occurred between first dose of study drug and up to 28 days after the last dose that were absent before treatment or worsened relative to pretreatment state. Grades of AEs were defined by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.03. Grade 1=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5= death related to AE.
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  All-causality TEAEs | 60
  All-causality Grade 3 or 4 TEAEs | 29
  All-causality Grade 5 TEAEs | 0
  Treatment-related TEAEs | 58
  Treatment-related Grade 3 or 4 TEAEs | 27
  Treatment-related Grade 5 TEAEs | 0

17. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Treatment-related SAEs were determined by the investigator.
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  All-causality SAEs | 11
  Treatment-related SAEs | 9

18. Secondary Outcome: Number of Participants With TEAEs Leading to Permanent Discontinuation of Study Drug
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. TEAEs were AEs that occurred between first dose of study drug and up to 28 days after the last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  All-causality TEAEs | 3
  Treatment-related TEAEs | 3

19. Secondary Outcome: Number of Participants With TEAEs Leading to Temporary Discontinuation of Study Drug
Description: as for outcome 18
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  All-causality TEAEs | 20
  Treatment-related TEAEs | 19

20. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Reduction of Study Drug
Description: as for outcome 18
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  All-causality TEAEs | 24
  Treatment-related TEAEs | 24

21. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory parameters included hematology, serum chemistry, urinalysis and coagulation. Grades of laboratory abnormalities were defined according to NCI CTCAE version 4.03. Participants with laboratory test abnormalities meeting specified criteria (>upper limit of normal [ULN] or <lower limit of normal [LLN]) (without regards to baseline abnormality) are reported.
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib. Number of participants analyzed refers to number of participants evaluable for this outcome measure. Number analyzed refers to total number of participants with at least 1 observation of the given laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  Erythrocyte Mean Corpuscular Volume <LLN | 1
  Erythrocyte Mean Corpuscular Volume >ULN | 33
  Erythrocytes <LLN: number analyzed (Participants) | 44
  Erythrocytes <LLN | 38
  Hematocrit <LLN | 39
  Blood urea nitrogen >ULN | 3
  Lactate dehydrogenase >ULN | 8
  Protein <LLN | 5
  Protein >ULN | 2
  Prothrombin Time <LLN: number analyzed (Participants) | 35
  Prothrombin Time <LLN | 2

22. Secondary Outcome: Number of Participants With Hematology Laboratory Results From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline
Description: Hematology laboratory parameters included hematocrit, hemoglobin, mean corpuscular volume, red blood cells, platelets, white blood cells with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils). Grades of lab results were defined by NCI CTCAE version 4.03. Grade 1(mild)=asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2(moderate)=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=life-threatening consequences, urgent intervention indicated; Grade 5=death related to AE. This outcome measure was based only on laboratory data. As Grade 4 anemia cannot be assessed based only on laboratory data, it was not applicable for analysis in this outcome measure.
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib. Number of participants analyzed refers to number of participants evaluable for this outcome measure. Number analyzed refers to total number of participants who had on-study laboratory test values that were applicable for the assessment of the laboratory results of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  Anemia Grade 0 to Grade 3 | 7
  Anemia Grade 1 to Grade 3 | 1
  Anemia Grade 2 to Grade 3 | 0
  Anemia Grade 0 to Grade 4: number analyzed (Participants) | 0
  Anemia Grade 1 to Grade 4: number analyzed (Participants) | 0
  Anemia Grade 2 to Grade 4: number analyzed (Participants) | 0
  Lymphocyte count decreased Grade 0 to Grade 3 | 1
  Lymphocyte count decreased Grade 1 to Grade 3 | 0
  Lymphocyte count decreased Grade 2 to Grade 3 | 0
  Lymphocyte count decreased Grade 0 to Grade 4 | 0
  Lymphocyte count decreased Grade 1 to Grade 4 | 0
  Lymphocyte count decreased Grade 2 to Grade 4 | 0
  Neutrophil count decreased Grade 0 to Grade 3 | 3
  Neutrophil count decreased Grade 0 to Grade 4 | 0
  Neutrophil count decreased Grade 1 to Grade 3 | 0
  Neutrophil count decreased Grade 1 to Grade 4 | 0
  Neutrophil count decreased Grade 2 to Grade 3 | 0
  Neutrophil count decreased Grade 2 to Grade 4 | 0
  White blood cell decreased Grade 0 to Grade 3 | 1
  White blood cell decreased Grade 0 to Grade 4 | 0
  White blood cell decreased Grade 1 to Grade 3 | 0
  White blood cell decreased Grade 1 to Grade 4 | 0
  White blood cell decreased Grade 2 to Grade 3 | 0
  White blood cell decreased Grade 2 to Grade 4 | 0

23. Secondary Outcome: Number of Participants With Chemistry Laboratory Results From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline
Description: Chemistry laboratory parameters included albumin, total protein, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, total bilirubin, blood urea nitrogen, creatinine, non-fasting glucose, bicarbonate, calcium, chloride, magnesium, phosphate, potassium, sodium, and lactate dehydrogenase. Grades of laboratory results were defined by NCI CTCAE version 4.03. Grade 1 (Mild) = asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2 (Moderate ) = minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3 = severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4 = events with life-threatening consequences, urgent intervention indicated; Grade 5 = death related to AE.
Time Frame: Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months)
Population: The analysis population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
Participants
  Hyperglycemia Baseline grade not reported to Grade 3 | 0
  Hyperglycemia Baseline grade not reported to Grade 4 | 0
  Hyperglycemia Grade 0 to Grade 3 | 1
  Hyperglycemia Grade 0 to Grade 4 | 0
  Hyperglycemia Grade 1 to Grade 3 | 0
  Hyperglycemia Grade 1 to Grade 4 | 0
  Hyperglycemia Grade 2 to Grade 3 | 0
  Hyperglycemia Grade 2 to Grade 4 | 0
  Hypophosphatemia Baseline grade not reported to Grade 3 | 0
  Hypophosphatemia Baseline grade not reported to Grade 4 | 0
  Hypophosphatemia Grade 0 to Grade 3 | 1
  Hypophosphatemia Grade 0 to Grade 4 | 0
  Hypophosphatemia Grade 1 to Grade 3 | 0
  Hypophosphatemia Grade 1 to Grade 4 | 0
  Hypophosphatemia Grade 2 to Grade 3 | 0
  Hypophosphatemia Grade 2 to Grade 4 | 0

24. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Talazoparib in Cycles 2, 3 and 4 in PK Analysis Set
Time Frame: Pre-dose on Day 1 of Cycles 2, 3, 4
Population: The analysis population included all participants treated with talazoparib with drug plasma concentration results from at least 1 visit. Number of participants analyzed=number of participants evaluable for this outcome measure. Number analyzed=number of participants evaluable for each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
picograms per milliliter (pg/mL)
  Cycle 2: number analyzed (Participants) | 58
  Cycle 2 | 4703 (71.5)
  Cycle 3: number analyzed (Participants) | 56
  Cycle 3 | 4699 (119.9)
  Cycle 4: number analyzed (Participants) | 58
  Cycle 4 | 4198 (139.8)

25. Secondary Outcome: Within-Participant Average Ctrough of Talazoparib at Steady State in PK Analysis Set
Description: Within-participant average Ctrough of talazoparib at steady state for each participant was defined as the average (mean) value of the steady state Ctrough values (Cycle 2 Day 1, Cycle 3 Day 1 and Cycle 4 Day 1 trough concentrations) for each individual participant.
Time Frame: Pre-dose on Day 1 of Cycles 2, 3, 4
Population: The analysis population included all participants treated with talazoparib for whom drug plasma concentration results from at least 1 visit were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 61
pg/mL | 4525 (109.5)

26. Secondary Outcome: Ctrough of Talazoparib in Cycles 2, 3 and 4 in Dose-Compliant PK Analysis Set
Time Frame: Pre-dose on Day 1 of Cycles 2, 3, 4
Population: The analysis population included all participants treated with talazoparib with drug plasma concentration results from at least 1 visit who had received 21 consecutive days of dosing without interruption prior to sample collection. Actual sample collection times were used to determine whether a pre-dose PK sample was dose-compliant. Number of participants analyzed=number of participants evaluable for this outcome measure. Number analyzed=number of participants evaluable for each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
pg/mL
  Cycle 2: number analyzed (Participants) | 41
  Cycle 2 | 5241 (57.9)
  Cycle 3: number analyzed (Participants) | 34
  Cycle 3 | 5208 (53.8)
  Cycle 4: number analyzed (Participants) | 34
  Cycle 4 | 4537 (84.6)

27. Secondary Outcome: Within-Participant Average Ctrough of Talazoparib at Steady State in Dose-Compliant PK Analysis Set
Description: as for outcome 25
Time Frame: Pre-dosing on Day 1 of Cycles 2, 3, 4
Population: The analysis population included all participants treated with talazoparib with drug plasma concentration results from at least 1 visit who had received 21 consecutive days of dosing without interruption prior to sample collection. Actual sample collection times were used to determine whether a pre-dose PK sample was dose-compliant.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
pg/mL | 5001 (65.2)

28. Secondary Outcome: Number of Participants Who Achieved Definitive Deterioration in Global Health Status (GHS)/Quality of Life (QoL) Per European Organization For Research And Treatment Of Cancer Quality Of Life Questionnaire (EORTC QLQ-30)
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes (PROs), consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the GHS/QoL scale, participants rated their overall health and quality of life within the past week. A 10 point change from baseline was used to indicate clinically meaningful change. Definitive deterioration was defined as ≥10 point decrease from baseline without any subsequent <10 point decrease.
Time Frame: Baseline to End of Treatment visit (assessed for maximum of 33 weeks)
Population: The analysis population included all participants who completed a baseline and at least 1 post-baseline QoL assessment prior to the end of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Participants | 19

29. Secondary Outcome: Kaplan-Meier Estimate of Time to Definitive Deterioration in GHS/QoL Per EORTC QLQ-30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the GHS/QoL scale, participants rated their overall health and quality of life within the past week. A 10 point change from baseline was used to indicate clinically meaningful change. Definitive deterioration was defined as ≥10 point decrease from baseline without any subsequent <10 point decrease.
Time Frame: Baseline to End of Treatment visit (assessed for maximum of 33 weeks)
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Months | NA [4.6 to NA] — The median time to definitive deterioration in GHS/QoL and the upper limit of its 95% confidence interval were not estimable as there was insufficient number of participants with definitive deterioration.

30. Secondary Outcome: Probability of Not Achieving Definitive Deterioration in GHS/QoL Per EORTC QLQ-C30 at 3 and 6 Months
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all to 4=very much).
  For the GHS/QoL scale, participants rated their overall health and quality of life within the past week. A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best. A 10 point change from baseline was used to indicate clinically meaningful change. Definitive deterioration was defined as ≥10 point decrease from baseline without any subsequent <10 point decrease.
  Probability of not achieving definitive deterioration (being event-free) at specified time points (3 and 6 months post-baseline) using the Kaplan Meier method were reported.
Time Frame: 3 months and 6 months post-baseline
Population: as for outcome 28
Measure: Number (95% Confidence Interval); unit: Probability of being event-free
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Probability of being event-free
  3 months | 0.696 [0.547 to 0.805]
  6 months | 0.594 [0.435 to 0.721]

31. Secondary Outcome: Number of Participants Who Achieved Definitive Deterioration in Nausea and Vomiting Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the nausea and vomiting symptoms scale, participants self-rated how much they had felt nauseated and/or vomited during the past week. A 10 point change from baseline was used to indicate clinically meaningful change. Definitive deterioration was defined as ≥10 point increase from baseline without any subsequent <10 point increase.
Time Frame: Baseline to End of Treatment visit (assessed for maximum of 33 weeks)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Participants | 9

32. Secondary Outcome: Kaplan-Meier Estimate of Time to Definitive Deterioration in Nausea and Vomiting Symptoms Per EORTC QLQ-C30
Description: as for outcome 31
Time Frame: Baseline to End of Treatment visit (assessed for maximum of 33 weeks)
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Months | NA [NA to NA] — The median time to definitive deterioration in nausea and vomiting symptoms and its 95% confidence interval were not estimable as there was insufficient number of participants with definitive deterioration.

33. Secondary Outcome: Probability of Not Achieving Definitive Deterioration in Nausea and Vomiting Symptoms Per EORTC QLQ-C30 at 3 and 6 Months
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, with 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores (1=very poor to 7=excellent); other items have 4 possible scores (1=not at all to 4=very much).
  For the nausea and vomiting symptoms scale, participants self-rated how much they had felt nauseated and/or vomited during the past week. A linear transformation was applied to raw scores so that transformed scores lie between 0 to 100, with 0 being the best and 100 being the worst for this symptom scale. A 10 point change from baseline was used to indicate clinically meaningful change. Definitive deterioration was defined as≥10 point increase from baseline without any subsequent <10 point increase. Probability of not achieving definitive deterioration (being event-free) at specified time points (3 and 6 months post-baseline) using Kaplan Meier method were reported.
Time Frame: 3 months and 6 months post-baseline
Population: as for outcome 28
Measure: Number (95% Confidence Interval); unit: Probability of being event-free
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Probability of being event-free
  3 months | 0.863 [0.734 to 0.932]
  6 months | 0.818 [0.678 to 0.901]

34. Secondary Outcome: Change From Baseline in Global QoL Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the GHS/QoL scale, participants rated their overall health and quality of life within the past week. Negative change from baseline indicates deterioration in GHS/QoL and positive change indicates improvement.
Time Frame: Baseline, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Day 1 of Cycles 3-6, End of Treatment visit (maximum of 33 weeks) and Post-surgical follow-up visit (maximum of 41 weeks)
Population: Number of Participants Analyzed refers to participants who completed the PRO assessment of this outcome measure at baseline and had at least 1 post-baseline assessment of this outcome measure prior to end of study treatment. Number Analyzed refers to those who completed the PRO assessment of this outcome measure at both baseline and each specific visit. "Number Analyzed" may or may not be smaller than "Number of participants analyzed" due to individual missing values.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -6.0 [-10.43 to -1.59]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -7.4 [-11.98 to -2.87]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -5.3 [-9.36 to -1.25]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -9.1 [-14.70 to -3.42]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -10.3 [-15.14 to -5.40]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | -13.0 [-19.29 to -6.78]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -11.3 [-17.17 to -5.41]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | -7.9 [-13.00 to -2.71]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | -13.3 [-19.64 to -7.02]

35. Secondary Outcome: Change From Baseline in Physical Functioning Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the physical functioning scale, participants self-rated levels of difficulty in doing strenuous activities, taking a walk, how much they needed to stay in bed or a chair, or needed help with eating, dressing, bathing, using the toilet. Negative change from baseline indicates deterioration in physical functioning and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -3.6 [-5.73 to -1.40]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -6.1 [-9.12 to -3.05]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -6.1 [-8.95 to -3.17]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -8.4 [-12.53 to -4.29]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -9.3 [-12.66 to -5.95]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | -9.7 [-14.39 to -5.10]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -9.0 [-13.82 to -4.24]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | -5.1 [-8.83 to -1.45]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | -14.2 [-21.16 to -7.28]

36. Secondary Outcome: Change From Baseline in Role Functioning Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the role functioning scale, participants self-rated how much they were limited in doing work or daily activities, or in pursuing hobbies or other leisure time activities during the past week. Negative change from baseline values indicates deterioration in role functioning and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -4.7 [-9.31 to 0.01]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -9.4 [-14.71 to -4.14]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -6.4 [-10.97 to -1.91]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -10.9 [-18.04 to -3.70]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -8.9 [-13.15 to -4.67]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | -9.4 [-15.94 to -2.87]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -7.0 [-12.85 to -1.13]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | -4.8 [-10.90 to 1.38]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | -21.7 [-31.49 to -11.84]

37. Secondary Outcome: Change From Baseline in Emotional Functioning Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the emotional functioning scale, participants self-rated how much they felt tense, worried, irritable or depressed during the past week. Negative change from baseline values indicates deterioration in emotional functioning and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 2.9 [-2.10 to 7.91]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 0.4 [-4.39 to 5.11]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 1.3 [-3.74 to 6.39]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -0.9 [-6.05 to 4.24]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -4.8 [-9.47 to -0.22]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | -3.0 [-8.89 to 2.90]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -7.8 [-14.54 to -1.06]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | -4.0 [-9.87 to 1.78]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | -3.1 [-10.61 to 4.50]

38. Secondary Outcome: Change From Baseline in Cognitive Functioning Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the cognitive functioning scale, participants self-rated the extent of difficulty in concentrating on things or remembering things during the past week. Negative change from baseline values indicates deterioration in cognitive functioning and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -2.3 [-7.02 to 2.37]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -5.4 [-9.62 to -1.25]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -5.3 [-9.78 to -0.83]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -6.9 [-12.93 to -0.84]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -9.7 [-15.64 to -3.74]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | -7.7 [-13.49 to -1.90]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -9.7 [-17.69 to -1.66]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | -7.1 [-13.84 to -0.44]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | -7.8 [-16.98 to 1.43]

39. Secondary Outcome: Change From Baseline in Social Functioning Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the social functioning scale, participants self-rated how much their physical condition or medical treatment interfered with their family life and social activities during the past week. Negative change from baseline values indicates deterioration in social functioning and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -2.3 [-8.62 to 3.96]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -4.3 [-9.71 to 1.02]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -1.9 [-7.16 to 3.37]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -7.6 [-14.18 to -1.03]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -5.4 [-10.00 to -0.85]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | -6.0 [-14.25 to 2.28]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -8.1 [-15.45 to -0.68]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | -8.1 [-14.21 to -1.98]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | -20.6 [-30.59 to -10.52]

40. Secondary Outcome: Change From Baseline in Fatigue Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the fatigue symptoms scale, participants self-rated how much they had felt weak, tired or needed to rest during the past week. Negative change from baseline values indicates improvement of fatigue symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 16.3 [9.98 to 22.58]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 18.4 [12.70 to 24.02]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 17.4 [11.58 to 23.27]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 21.0 [13.88 to 28.15]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 22.2 [16.74 to 27.71]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 21.7 [14.45 to 28.85]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 20.4 [12.41 to 28.45]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 14.3 [7.32 to 21.25]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 23.3 [16.33 to 30.34]

41. Secondary Outcome: Change From Baseline in Nausea and Vomiting Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the nausea and vomiting symptoms scale, participants self-rated how much they had felt nauseated and/or vomited during the past week. Negative change from baseline values indicates improvement of nausea and vomiting symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 11.2 [6.80 to 15.68]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 8.0 [4.40 to 11.55]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 7.2 [3.67 to 10.72]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 5.4 [1.97 to 8.90]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 3.9 [0.74 to 7.01]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 4.3 [1.06 to 7.49]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 7.5 [2.83 to 12.22]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 0.5 [-2.46 to 3.42]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 1.1 [-2.13 to 4.35]

42. Secondary Outcome: Change From Baseline in Pain Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the pain symptoms scale, participants self-rated the extent of pain and how much the pain interfered with daily activities during the past week. Negative change from baseline values indicates improvement of pain symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -1.9 [-6.01 to 2.13]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -0.0 [-4.78 to 4.78]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -1.5 [-6.50 to 3.47]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 0.7 [-4.99 to 6.44]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -2.7 [-7.83 to 2.41]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 1.3 [-6.09 to 8.66]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -1.1 [-7.76 to 5.61]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 1.4 [-4.36 to 7.22]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 14.4 [6.65 to 22.24]

43. Secondary Outcome: Change From Baseline in Dyspnoea Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the dyspnoea symptoms scale, participants self-rated the intensity of shortness of breath during the past week. Negative change from baseline values indicates improvement of dyspnoea symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -0.8 [-2.34 to 0.79]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 5.1 [0.42 to 9.72]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 5.3 [0.44 to 10.16]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 8.0 [2.38 to 13.56]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 16.3 [9.43 to 23.13]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 8.5 [3.16 to 13.93]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 8.6 [2.31 to 14.89]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 3.8 [-0.81 to 8.43]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 4.4 [-2.67 to 11.56]

44. Secondary Outcome: Change From Baseline in Insomnia Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the insomnia symptoms scale, participants self-rated the intensity of shortness of breath during the past week. Negative change from baseline values indicates improvement of insomnia symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -4.7 [-12.59 to 3.29]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -4.3 [-13.10 to 4.41]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -10.6 [-18.72 to -2.49]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -6.5 [-14.50 to 1.46]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | -7.0 [-15.52 to 1.56]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | -2.6 [-12.90 to 7.77]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | -6.5 [-18.85 to 5.94]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | -4.8 [-16.59 to 7.07]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 1.1 [-13.68 to 15.90]

45. Secondary Outcome: Change From Baseline in Appetite Loss Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the appetite loss symptoms scale, participants self-rated the extent of lack of appetite during the past week. Negative change from baseline values indicates improvement of appetite loss symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 10.1 [2.47 to 17.68]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 3.6 [-3.37 to 10.62]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 0.8 [-6.32 to 7.84]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 5.8 [-2.63 to 14.22]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 3.1 [-3.91 to 10.11]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 4.3 [-3.64 to 12.18]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 4.3 [-4.48 to 13.09]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 1.9 [-4.87 to 8.67]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 2.2 [-5.74 to 10.18]

46. Secondary Outcome: Change From Baseline in Constipation Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the constipation symptoms scale, participants self-rated the intensity of constipation during the past week. Negative change from baseline values indicates improvement of constipation symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 12.4 [5.32 to 19.49]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 9.4 [1.71 to 17.13]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 12.1 [4.84 to 19.40]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 8.0 [0.69 to 15.26]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 6.2 [-0.23 to 12.63]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 7.7 [0.48 to 14.90]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 5.4 [-4.65 to 15.41]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 3.8 [-1.58 to 9.20]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 3.3 [-4.90 to 11.57]

47. Secondary Outcome: Change From Baseline in Diarrhea Symptoms Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the diarrhea symptoms scale, participants self-rated the intensity of diarrhea during the past week. Negative change from baseline values indicates improvement of diarrhea symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 1.6 [-2.30 to 5.40]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 2.2 [-1.68 to 6.02]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 1.5 [-2.24 to 5.27]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 0.0 [-2.09 to 2.09]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 2.3 [-1.14 to 5.79]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 3.4 [-1.41 to 8.25]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 0.0 [-4.46 to 4.46]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 1.9 [-0.79 to 4.60]
  Post--surgical follow-up: number analyzed (Participants) | 30
  Post--surgical follow-up | 1.1 [-2.87 to 5.09]

48. Secondary Outcome: Change From Baseline in Financial Difficulties Per EORTC QLQ-C30
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the symptom scale of financial difficulties, participants self-rated how much their physical condition or medical treatment caused financial difficulties. Negative change from baseline values indicates improvement of financial difficulties and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Median (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 50
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -3.9 [-8.47 to 0.72]
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | -1.4 [-9.52 to 6.62]
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | -3.0 [-11.15 to 5.09]
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | -0.7 [-8.39 to 6.94]
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 1.6 [-6.81 to 9.91]
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 5.1 [-5.25 to 15.51]
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 3.2 [-8.31 to 14.76]
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 10.5 [-0.20 to 21.15]
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 16.7 [4.55 to 28.79]

49. Secondary Outcome: Change From Baseline in Body Image Per EORTC QLQ Breast Cancer Quality of Life Questionnaire (EORTC QLQ-BR23)
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the functional scale of body image, participants self-rated how much they felt physically less attractive or less feminine, difficult to look at themselves naked, or dissatisfied with their body during the past week. Negative change from baseline indicates worsening of self-rated body image and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 49
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 0.2 [-2.79 to 3.18]
  Cycle 2 Day 1: number analyzed (Participants) | 44
  Cycle 2 Day 1 | 1.7 [-1.37 to 4.78]
  Cycle 2 Day 15: number analyzed (Participants) | 43
  Cycle 2 Day 15 | -0.2 [-3.84 to 3.45]
  Cycle 3 Day 1: number analyzed (Participants) | 45
  Cycle 3 Day 1 | -0.4 [-3.53 to 2.79]
  Cycle 4 Day 1: number analyzed (Participants) | 42
  Cycle 4 Day 1 | -6.3 [-11.11 to -1.59]
  Cycle 5 Day 1: number analyzed (Participants) | 38
  Cycle 5 Day 1 | -9.4 [-15.17 to -3.69]
  Cycle 6 Day 1: number analyzed (Participants) | 30
  Cycle 6 Day 1 | -6.1 [-11.08 to -1.14]
  End of treatment: number analyzed (Participants) | 34
  End of treatment | -6.9 [-12.10 to -1.63]
  Post-surgical follow-up: number analyzed (Participants) | 29
  Post-surgical follow-up | -13.8 [-20.64 to -6.95]

50. Secondary Outcome: Change From Baseline in Sexual Functioning Per EORTC QLQ-BR23
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the sexual functioning scale, participants self-rated to what extent they were interested in sex and were sexually active (with or without intercourse) during the past 4 weeks. Negative change from baseline values indicates worsening of sexual functioning and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 49
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -1.6 [-7.45 to 4.35]
  Cycle 2 Day 1: number analyzed (Participants) | 44
  Cycle 2 Day 1 | -3.0 [-9.33 to 3.27]
  Cycle 2 Day 15: number analyzed (Participants) | 43
  Cycle 2 Day 15 | -2.7 [-8.73 to 3.31]
  Cycle 3 Day 1: number analyzed (Participants) | 45
  Cycle 3 Day 1 | -0.4 [-7.33 to 6.59]
  Cycle 4 Day 1: number analyzed (Participants) | 42
  Cycle 4 Day 1 | -1.2 [-8.39 to 6.01]
  Cycle 5 Day 1: number analyzed (Participants) | 38
  Cycle 5 Day 1 | -3.5 [-11.17 to 4.15]
  Cycle 6 Day 1: number analyzed (Participants) | 30
  Cycle 6 Day 1 | -2.8 [-11.59 to 6.04]
  End of treatment: number analyzed (Participants) | 34
  End of treatment | -3.4 [-11.11 to 4.25]
  Post-surgical follow-up: number analyzed (Participants) | 29
  Post-surgical follow-up | -10.9 [-20.55 to -1.29]

51. Secondary Outcome: Change From Baseline in Sexual Enjoyment Per EORTC QLQ-BR23
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the functional scale of sexual enjoyment, participants self-rated to what extent sex was enjoyable for them during the past 4 weeks. Negative change from baseline values indicates worsening of sexual enjoyment and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 26
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 20
  Cycle 1 Day 15 | -3.3 [-11.95 to 5.29]
  Cycle 2 Day 1: number analyzed (Participants) | 21
  Cycle 2 Day 1 | 0.0 [-11.75 to 11.75]
  Cycle 2 Day 15: number analyzed (Participants) | 18
  Cycle 2 Day 15 | -3.7 [-16.28 to 8.87]
  Cycle 3 Day 1: number analyzed (Participants) | 19
  Cycle 3 Day 1 | -10.5 [-21.31 to 0.25]
  Cycle 4 Day 1: number analyzed (Participants) | 19
  Cycle 4 Day 1 | -12.3 [-23.27 to -1.29]
  Cycle 5 Day 1: number analyzed (Participants) | 17
  Cycle 5 Day 1 | -5.9 [-18.35 to 6.59]
  Cycle 6 Day 1: number analyzed (Participants) | 13
  Cycle 6 Day 1 | -12.8 [-28.29 to 2.65]
  End of treatment: number analyzed (Participants) | 15
  End of treatment | -13.3 [-30.14 to 3.47]
  Post-surgical follow-up: number analyzed (Participants) | 9
  Post-surgical follow-up | -18.5 [-37.13 to 0.10]

52. Secondary Outcome: Change From Baseline in Future Perspective Per EORTC QLQ-BR23
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the functional scale of future perspective, participants self-rated how much they were worried about their health in the future. Negative change from baseline values indicates worsening of future perspective and positive change indicates improvement.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 49
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 3.1 [-3.91 to 10.11]
  Cycle 2 Day 1: number analyzed (Participants) | 44
  Cycle 2 Day 1 | 11.4 [3.50 to 19.23]
  Cycle 2 Day 15: number analyzed (Participants) | 43
  Cycle 2 Day 15 | 11.6 [3.91 to 19.34]
  Cycle 3 Day 1: number analyzed (Participants) | 45
  Cycle 3 Day 1 | 5.9 [-2.42 to 14.27]
  Cycle 4 Day 1: number analyzed (Participants) | 42
  Cycle 4 Day 1 | 5.6 [-2.36 to 13.48]
  Cycle 5 Day 1: number analyzed (Participants) | 38
  Cycle 5 Day 1 | 6.1 [-1.86 to 14.14]
  Cycle 6 Day 1: number analyzed (Participants) | 30
  Cycle 6 Day 1 | 6.7 [-3.87 to 17.21]
  End of treatment: number analyzed (Participants) | 34
  End of treatment | -2.0 [-12.26 to 8.34]
  Post-surgical follow-up: number analyzed (Participants) | 29
  Post-surgical follow-up | 10.3 [-0.95 to 21.64]

53. Secondary Outcome: Change From Baseline in Systemic Therapy Side Effects Per EORTC QLQ-BR23
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the systemic therapy side effects scale, participants self-rated the intensity of symptoms of dry mouth, unusual taste, pain and irritation of eyes, hair loss, feeling ill or unwell, hot flushes and headaches during the past week. Negative change from baseline= improvement of these side effects, positive change = deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 49
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 7.1 [3.74 to 10.43]
  Cycle 2 Day 1: number analyzed (Participants) | 44
  Cycle 2 Day 1 | 6.6 [3.70 to 9.50]
  Cycle 2 Day 15: number analyzed (Participants) | 43
  Cycle 2 Day 15 | 9.1 [5.90 to 12.26]
  Cycle 3 Day 1: number analyzed (Participants) | 45
  Cycle 3 Day 1 | 11.2 [7.57 to 14.87]
  Cycle 4 Day 1: number analyzed (Participants) | 42
  Cycle 4 Day 1 | 15.0 [10.93 to 19.00]
  Cycle 5 Day 1: number analyzed (Participants) | 38
  Cycle 5 Day 1 | 13.5 [9.10 to 17.97]
  Cycle 6 Day 1: number analyzed (Participants) | 30
  Cycle 6 Day 1 | 16.5 [11.57 to 21.44]
  End of treatment: number analyzed (Participants) | 34
  End of treatment | 6.9 [3.22 to 10.50]
  Post-surgical follow-up: number analyzed (Participants) | 29
  Post-surgical follow-up | 3.3 [-0.28 to 6.84]

54. Secondary Outcome: Change From Baseline in Breast Symptoms Per EORTC QLQ-BR23
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the breast symptoms scale, participants self-rated how much they had pain or skin problems (e.g. itchy, dry, flaky) on or in the area of affected breast, and how much this area was swollen or oversensitive during the past week. Negative change from baseline indicates improvement of breast symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 49
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -2.1 [-5.97 to 1.71]
  Cycle 2 Day 1: number analyzed (Participants) | 44
  Cycle 2 Day 1 | -4.9 [-9.02 to -0.82]
  Cycle 2 Day 15: number analyzed (Participants) | 43
  Cycle 2 Day 15 | -9.1 [-13.61 to -4.60]
  Cycle 3 Day 1: number analyzed (Participants) | 45
  Cycle 3 Day 1 | -8.0 [-12.20 to -3.73]
  Cycle 4 Day 1: number analyzed (Participants) | 42
  Cycle 4 Day 1 | -5.6 [-9.72 to -1.39]
  Cycle 5 Day 1: number analyzed (Participants) | 38
  Cycle 5 Day 1 | -7.7 [-12.75 to -2.61]
  Cycle 6 Day 1: number analyzed (Participants) | 30
  Cycle 6 Day 1 | -6.4 [-11.85 to -0.93]
  End of treatment: number analyzed (Participants) | 34
  End of treatment | 0.2 [-5.55 to 6.04]
  Post-surgical follow-up: number analyzed (Participants) | 29
  Post-surgical follow-up | 8.6 [-0.16 to 17.40]

55. Secondary Outcome: Change From Baseline in Arm Symptoms Per EORTC QLQ-BR23
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the arm symptoms scale, participants self-rated how much they had pain in the arm or shoulder, how much the arm or hand was swollen, and difficulty in raising the arm or moving it sideways. Negative change from baseline indicates improvement of arm symptoms and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 49
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | -1.6 [-4.59 to 1.49]
  Cycle 2 Day 1: number analyzed (Participants) | 44
  Cycle 2 Day 1 | -0.8 [-4.05 to 2.53]
  Cycle 2 Day 15: number analyzed (Participants) | 43
  Cycle 2 Day 15 | -1.6 [-5.25 to 2.15]
  Cycle 3 Day 1: number analyzed (Participants) | 45
  Cycle 3 Day 1 | -0.7 [-4.40 to 2.92]
  Cycle 4 Day 1: number analyzed (Participants) | 42
  Cycle 4 Day 1 | -1.3 [-4.40 to 1.76]
  Cycle 5 Day 1: number analyzed (Participants) | 38
  Cycle 5 Day 1 | 0.3 [-3.73 to 4.32]
  Cycle 6 Day 1: number analyzed (Participants) | 30
  Cycle 6 Day 1 | -1.5 [-6.20 to 3.23]
  End of treatment: number analyzed (Participants) | 34
  End of treatment | -1.0 [-5.18 to 3.22]
  Post-surgical follow-up: number analyzed (Participants) | 29
  Post-surgical follow-up | 13.0 [5.70 to 20.35]

56. Secondary Outcome: Change From Baseline in Upset by Hair Loss Per EORTC QLQ-BR23
Description: EORTC-QLQ-BR23 is a 23-item breast cancer module developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer, consisting of 2 functional scales, 3 symptoms scales, and 3 single-item scales. Each scale has 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for functional scales, and 0 being the best and 100 being the worst for symptoms scales.
  For the upset by hair loss scale, participants self-rated how upset they were due to loss of hair during the past week. Negative change from baseline values indicates improvement of upset by hair loss and positive change indicates deterioration.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 3
Units on a scale
  Cycle 1 Day 15: number analyzed (Participants) | 1
  Cycle 1 Day 15 | 0.0 [NA to NA] — 95% CI was not reported for n=1
  Cycle 2 Day 1: number analyzed (Participants) | 2
  Cycle 2 Day 1 | -33.3 [-456.87 to 390.21]
  Cycle 2 Day 15 | -11.1 [-137.60 to 115.37]
  Cycle 3 Day 1: number analyzed (Participants) | 2
  Cycle 3 Day 1 | 33.33 [33.33 to 33.33]
  Cycle 4 Day 1 | 11.1 [-161.26 to 183.48]
  Cycle 5 Day 1: number analyzed (Participants) | 0
  Cycle 6 Day 1: number analyzed (Participants) | 0
  End of treatment: number analyzed (Participants) | 1
  End of treatment | 33.33 [NA to NA] — 95% CI was not reported for n=1
  Post-surgical follow-up: number analyzed (Participants) | 1
  Post-surgical follow-up | 33.3 [NA to NA] — 95% CI was not reported for n=1

57. Secondary Outcome: Number of Participants With Deterioration in Nausea/Vomiting Symptoms
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales. For the nausea and vomiting symptoms scale, participants self-rated how much they had felt nauseated and/or vomited during the past week. A 10 point change from baseline was used to indicate clinically meaningful change. Deterioration in nausea and vomiting symptoms was defined as a 10 point or more increase from baseline for that specific time point.
Time Frame: as for outcome 34
Population: The analysis population included all participants who completed a baseline and at least one post-baseline QoL assessment prior to end of study treatment. Number of Participants Analyzed refers to participants who were evaluable for this outcome measure. Number analyzed refers to participants who were evaluable for this outcome measure at the specific visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Participants
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 21
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 20
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 18
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 14
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 10
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 11
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 10
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 3
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 5

58. Secondary Outcome: Number of Participants With Improvement in Nausea/Vomiting Symptoms
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales. For the nausea and vomiting symptoms scale, participants self-rated how much they had felt nauseated and/or vomited during the past week. A 10 point change from baseline was used to indicate clinically meaningful change. Improvement in nausea and vomiting symptoms was defined as a 10 point or more decrease from baseline for that specific time point.
Time Frame: as for outcome 34
Population: as for outcome 57
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Participants
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 1
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 2
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 2
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 2
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 2
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 2
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 0
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 3
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 3

59. Secondary Outcome: Number of Participants With No Change in Nausea/Vomiting Symptoms
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a GHS/QoL scale, and 6 single-item scales. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all to 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for GHS/QoL and functional scales, and 0 being the best and 100 being the worst for symptoms scales. For the nausea and vomiting symptoms scale, participants self-rated how much they had felt nauseated and/or vomited during the past week. A 10 point change from baseline was used to indicate clinically meaningful change. No change in nausea/vomiting symptoms=having neither deterioration (≥10 point increase from baseline) nor improvement (≥10 point decrease from baseline) for the time point.
Time Frame: as for outcome 34
Population: as for outcome 57
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 51
Participants
  Cycle 1 Day 15: number analyzed (Participants) | 43
  Cycle 1 Day 15 | 21
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 24
  Cycle 2 Day 15: number analyzed (Participants) | 44
  Cycle 2 Day 15 | 24
  Cycle 3 Day 1: number analyzed (Participants) | 46
  Cycle 3 Day 1 | 30
  Cycle 4 Day 1: number analyzed (Participants) | 43
  Cycle 4 Day 1 | 31
  Cycle 5 Day 1: number analyzed (Participants) | 39
  Cycle 5 Day 1 | 26
  Cycle 6 Day 1: number analyzed (Participants) | 31
  Cycle 6 Day 1 | 21
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 29
  Post-surgical follow-up: number analyzed (Participants) | 30
  Post-surgical follow-up | 22

60. Secondary Outcome: Number of Participants With Missed Expected Menstrual Periods Per Patient Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: Missed expected menstrual period was assessed electronically using the PRO CTCAE questionnaire, a PRO measure developed to evaluate symptomatic toxicity in patients on cancer clinical trials. This objective captures the concept of fertility preservation through PRO, since there is a possible fertility sparing effect of talazoparib versus chemotherapy.
Time Frame: as for outcome 34
Population: The analysis population included all participants who completed a baseline and at least 1 post-baseline QoL assessment prior to the end of the study treatment. Post-menopausal participants were excluded from this evaluation. Number of participants analyzed refers to the number of participants who were evaluable for this outcome measure. Number analyzed refers to the number of participants evaluable for each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 32
Participants
  Baseline: number analyzed (Participants) | 30
  Baseline | 0
  Cycle 1 Day 15: number analyzed (Participants) | 24
  Cycle 1 Day 15 | 1
  Cycle 2 Day 1: number analyzed (Participants) | 27
  Cycle 2 Day 1 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 27
  Cycle 2 Day 15 | 2
  Cycle 3 Day 1: number analyzed (Participants) | 30
  Cycle 3 Day 1 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 26
  Cycle 4 Day 1 | 3
  Cycle 5 Day 1: number analyzed (Participants) | 23
  Cycle 5 Day 1 | 1
  Cycle 6 Day 1: number analyzed (Participants) | 18
  Cycle 6 Day 1 | 1
  End of treatment: number analyzed (Participants) | 19
  End of treatment | 0
  Post-surgical follow-up: number analyzed (Participants) | 15
  Post-surgical follow-up | 1

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from Baseline to 28 days after the last dose of talazoparib (maximum of approximately 8 months). All-cause mortality was assessed from Baseline until participant died or withdrew consent for follow-up, or study termination (maximum of approximately 16 months).
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Talazoparib 1 mg QD
All-Cause Mortality (participants affected / at risk) | 2/61
Serious Adverse Events (participants affected / at risk) | 11/61
Other Adverse Events (participants affected / at risk) | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 1 mg QD (N=61)
Anaemia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 1 mg QD (N=61)
Anaemia (Blood and lymphatic system disorders) | 30
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 13
Dry mouth (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 42
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 48
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 7
Neutrophil count decreased (Investigations) | 9
White blood cell count decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 20
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 26
Anxiety (Psychiatric disorders) | 11
Insomnia (Psychiatric disorders) | 11
Breast pain (Reproductive system and breast disorders) | 7
Menstruation irregular (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 35
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 7
Hot flush (Vascular disorders) | 7
Hypertension (Vascular disorders) | 6

LIMITATIONS AND CAVEATS:
The study was prematurely terminated by the sponsor due to a change in clinical development strategy not related to safety or efficacy after all participants completed safety follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT03499353/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT03499353/SAP_001.pdf